CLINICAL TRIAL: NCT06389916
Title: Euclid Phoenix Lens Design Trial Phase 1
Brief Title: Euclid Phoenix Lens Design Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Euclid Systems Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EU-PHX-RCT-001
Record Dates: First submitted 2023-10-31; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Myopia; Cornea
MeSH Terms: conditions — Myopia; Corneal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Euclid orthokeratology MAX (current design) (Experimental): Euclid Orthokeratology (oprifocon A) Contact Lenses are lathe cut contact lenses with spherical posterior surfaces. The posterior curve is selected to properly fit an individual eye for orthokeratology and the anterior curve is selected to provide the necessary optical power for a temporary reduction of myopia. A peripheral curve system on the posterior surface allows tear exchange between the lens and the cornea.
  Interventions: Device: Euclid orthokeratology MAX (current design)
- Euclid orthokeratology MAX Phoenix (new design) (Experimental): Euclid Orthokeratology (oprifocon A) Contact Lenses are lathe cut contact lenses with spherical posterior surfaces. The posterior curve is selected to properly fit an individual eye for orthokeratology and the anterior curve is selected to provide the necessary optical power for a temporary reduction of myopia. A peripheral curve system on the posterior surface allows tear exchange between the lens and the cornea.
  Interventions: Device: Euclid orthokeratology MAX Phoenix (new design)

INTERVENTIONS:
Device: Euclid orthokeratology MAX (current design) — The current lens design
  Arms: Euclid orthokeratology MAX (current design)
Device: Euclid orthokeratology MAX Phoenix (new design) — The new lens design
  Arms: Euclid orthokeratology MAX Phoenix (new design)

SUMMARY:
The "first fit" success rate of the current Euclid orthokeratology "MAX" lens design will be compared to that of the new Euclid orthokeratology MAX "Phoenix" lens design in 30 children.

DETAILED DESCRIPTION:
The primary objective of this trial is to provide an assessment of the "first fit" success of the Euclid orthokeratology "Phoenix" lens design versus its current "MAX" lens design when used by practitioners with moderate experience with fitting Euclid MAX orthokeratology lenses.

The hypothesis to be tested is that the "first fit" success of the redesign Euclid MAX "Phoenix" lens design is greater than that of the current MAX lens design.

The primary outcome variable is the percentage of participants successfully fit with the first lenses empirically ordered for the existing MAX lens design versus a modified MAX lens ("Phoenix") design.

This clinical investigation will be a prospective, randomized, double-masked two-arm non-crossover trial.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age or, if under legal age have written consent of their parent or guardian to participate.
* Sign written Informed Consent (and the California Bill of Rights, if applicable).
* Ages 6-18 (inclusive) and able to understand and assent to participation
* Have need of optical correction for myopia, from -1.00 to -5.00 dioptcrs (D).
* Have a refractive astigmatism of less than -1.50 D.
* Have a minimum Best Spectacle Corrected Visual Acuity (BSCVA) of 20/40 or better.
* Have reasonable expectations of improvement in visual acuity with the Euclid Orthokeratology Lens of 20/40 or better after overnight wear without corrective aids.
* Be at least 18 years old to give informed consent.
* Not a current or former wearer of orthokeratology lenses
* Not a current wearer of soft contact lenses
* Have acceptable or optimal fit with study lenses and be willing to wear these lenses as directed for the duration of the study.
* On examination, have ocular findings considered to be within normal limits
* Normal binocularity (no amblyopia or strabismus, and no anisometropia of greater than 2.00D)
* Be willing and able to follow instructions and attend the schedule of follow-up visits.

Exclusion Criteria:

* Does not meet the any of the above inclusion criteria
* Not able or willing to provide informed consent and assent
* Requires concurrent ocular medication
* Eye injury or surgery within twelve weeks immediately prior to enrollment
* Pre-existing ocular condition that would preclude contact lens fitting
* Currently enrolled in an ophthalmic clinical trial
* Pregnant or lactating or expect to become pregnant during the trial
* Evidence of systemic or ocular abnormality, infection or disease likely to affect successful wear of contact lenses or use of their accessory solutions.
* Allergy or sensitivity to any product used in this trial
* Any systemic disease including autoimmune disease, immunocompromising diseases, connective tissue disease, clinically significant atopic diseases, insulin dependent diabetes, use of medications including corticosteroids and antimetabolites that may affect the eye or be exaggerated by contact lenses.
* Strabismus/amblyopia
* Habitually uncorrected anisometropia ≥2.00
* Subjects who have undergone corneal refractive surgery
* Subjects with severe corneal irregularity contraindicating lens wear
* Inability to wear contact lenses, or an unacceptable contact lens fit
* Poor or unacceptable fit with any study lens

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
First fit success rate | 1 month
  Percentage of children successfully fit in the first lens pair ordered (as determined by the PI)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Insight Vision Center Optometry, Costa Mesa, California
  - Dau Family Eye Care, Saint Johns, Florida
  - Cornea and Contact Lens Institute of Minnesota, Edina, Minnesota
  - Somerset Eye Care, North Brunswick, New Jersey
  - Treehouse Eyes, Tysons Corner, Virginia

IPD SHARING:
Plan to Share IPD: Undecided